CLINICAL TRIAL: NCT06803056
Title: QUANTIFY: Quantitative Understanding of Advanced Novel Techniques for Imaging Fasciitis and Yielding Biomarkers
Acronym: QUANTIFY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruth Chimenti (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Rochester Institute of Technology (Other)
Responsible Party: Sponsor-Investigator, Ruth Chimenti, Assistant Professor, Physical Therapy and Rehabilitation Science, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202409110; R61AT012275 (NIH)
Record Dates: First submitted 2024-12-12; First posted 2025-01-31 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Plantar Fasciopathy; Achilles Tendinopathy; Controls
Keywords: plantar fasciitis; achilles tendinitis; biomarker; myofascial; magnetic resonance imaging; ultrasound imaging; pain
MeSH Terms: conditions — Fasciitis, Plantar; Pain | interventions — Ultrasonography; Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: All participants will complete a clinical exam of the foot and ankle to identify painful myofascial tissue. All participants will subsequently have magnetic resonance imaging and ultrasound imaging of their foot and ankle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Diagnostic imaging (Other): All participants will have a clinical exam, magnetic resonance imaging, and ultrasound imaging of their foot and ankle.
  Interventions: Diagnostic Test: Clinical exam; Diagnostic Test: Ultrasound imaging; Diagnostic Test: Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Clinical exam — An experienced physical therapist with expertise in dry needling will confirm study eligibility and complete a standard clinical exam for myofascial pain. Gold standard for diagnosing myofascial pain as defined by Travell and Simons will be used. The criteria for muscle trigger point (TrP) include: 1) a taut band of skeletal muscle that is tender to palpation, 2) sustained compression of the taut band reproduces or exacerbates the participant's symptoms. Healthy tissue is defined as no palpable taut band.
Diagnostic Test: Ultrasound imaging — Shear wave elastography and b-mode ultrasound imaging techniques will capture the biomechanical and structural profile of foot and ankle muscle on the involved side.
Diagnostic Test: Magnetic Resonance Imaging — T1rho and IDEAL sequences will be used to capture the biochemical and structural profile of foot and ankle muscles on the involved side

SUMMARY:
This study is to create a test that can accurately find and measure the problem areas in muscle and fascia tissue, also known as myofascial pain. The hypothesis is that a combination of imaging findings will be able to detect when myofascial pain is present. The goal is to improve management of myofascial pain by making better tools to find changes in the muscle and fascia tissues for a more personalized treatment. This project was funded by the HEAL initiative (https://heal.nih.gov/).

DETAILED DESCRIPTION:
The objective of the R61 phase is to use novel imaging techniques to develop a diagnostic biosignature to objectively and accurately determine the location and severity of abnormal myofascial tissue. A cross-sectional study design approach with 3 groups: plantar fasciitis (n=50), Achilles tendinopathy (n=25), and pain-free controls (n=25) to test Specific Aim: Develop a diagnostic imaging biosignature of myofascial tissue to differentiate individuals with plantar fasciitis from other foot pain without a myofascial component (Achilles tendinopathy) and from matched pain-free controls.

The goal is to develop a diagnostic imaging biosignature that will be able to distinguish between A-MTrP in individuals with plantar fasciitis compared to healthy tissue control (pain-free controls). The biosignature developed in this R61 phase will be screened for clinical utility and considered of interest for further study if it meets the following milestone criteria: area under the receiver operating characteristic curve (ROC AUC) >0.7, sensitivity >60%, and specificity >60%. The ROC analysis will estimate diagnostic performance by comparing differences in biosignatures between tissue where myofascial pain is present vs. tissue where pain is absent.

The proposed sample size of 50 individuals with plantar fasciitis, 25 individuals with Achilles tendinopathy, and 25 matched controls was chosen to provide a confidence interval halfwidth of 0.10 for an AUC of 0.70, assuming 5 muscle measurements for each participant and an overall A-MTrPs prevalence of 0.36 in individuals with plantar fasciitis. Further assuming the 20 biomarkers to be considered in the R61 phase have AUCs uniformly distributed from 0.5 to 0.8, will have at least 85% power to obtain a biosignature meeting the milestone criteria.

ELIGIBILITY:
Inclusion criteria for plantar fasciitis group:

* Clinical diagnosis of plantar fasciitis
* Duration of plantar fasciitis pain greater than or equal to 3 months
* Severity of plantar fasciitis pain greater than or equal to 3/10

Inclusion criteria for Achilles tendinopathy group:

* Clinical diagnosis of insertional Achilles tendinopathy:
* Duration of Achilles tendinopathy pain greater than or equal to 3 months
* Severity of Achilles tendon pain greater than or equal to 3/10

Control group:

• Similar age, sex, and BMI as plantar fasciitis and Achilles tendinopathy groups

Exclusion criteria:

* Younger than 18 years of age
* History of an invasive procedures to the foot and ankle on the side of interest
* History of lower extremity injections, dry needling, or EPAT/ESWT within past 3 months on the side of interest
* Contraindications for MRI (e.g. non-MR compatible implanted devices, claustrophobia, inability to remain still comfortably for 1 hour in a supine position, body size too large for MR scanner)
* Clinically unstable medical or psychiatric issues
* Pregnant or possibly pregnant
* Co-morbidities associated with changes in musculoskeletal imaging, including: Diagnosed systemic conditions affecting the foot and ankle (e.g., rheumatoid arthritis, spondyloarthropathy, gout) endocrine disorder with complications (e.g., uncontrolled Type I or II diabetes, diabetic peripheral neuropathy) Neuromuscular diseases (e.g., Charcot-Marie-Tooth (CMT) disease) Connective tissue disorder (e.g. Marfan's syndrome, Ehlers-Danlos) Osteoarthritis of the foot or ankle History of foot or ankle fracture Infection of the foot or ankle (e.g., infectious fasciitis, calcaneal osteomyelitis) within the past year Familial hypercholesterolemia Neoplasms involving the foot, Plantar fibromatosis
* Control group only: Persistent or recurrent leg pain in the past 6 months
* Plantar fasciitis and Achilles tendinopathy groups only: Other source of heel or foot pain (e.g., tarsal tunnel syndrome, peripheral neuropathy, lumbar radiculopathy, calcaneal stress fracture, Morton's neuroma, fibromyalgia) or co-occurring plantar fasciitis and Achilles tendinopathy (for the Achilles tendinopathy group).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Reference Test: Trigger point (TrP) | Enrollment
  Travell and Simons' criteria will be used to identify active muscle trigger points (TrPs) as present or absent. The score will be "Yes" for present and "No" for absent.
Diagnostic Index Test: Imaging biosignature | Enrollment
  The biosignature will include a combination of ultrasound and/or magnetic resonance imaging measures to capture biomechanical, biochemical, and structural profile of myofascial tissue. Current key candidate imaging biomarkers include: T1p of muscle and fascia, Elastic modulus of the muscle, Shear strain of the plantar fascia, Fat fraction of the muscle, and Thickness of the plantar fascia. The is currently no established scale for this biosignature, which will be developed as part of this study.

SECONDARY OUTCOMES:
Pain Intensity and Interference | Enrollment
  The PEG (Pain, Enjoyment, General activity) is a three-item scale to assess pain intensity and interference. Each question is rated from 0 (least) to 10 (worst) and the scores are averaged to calculate a total PEG score.
Movement-evoked pain | Enrollment
  Participants will rate their pain using a verbal numeric rating scale (0-10) during walking where "0" represents "no pain" and "10" represents "worst pain imaginable"
Physical Function | Enrollment
  Participants will report their level of physical function using the PROMIS (Patient-Reported Outcomes Measurement Information System) Physical Function, Short form 6b. For PROMIS measures the general population mean is 50 with a standard deviation of 10. Impaired physical function would be indicated by a score less than 40.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Sluka, PT, PhD, Principal Investigator — University of Iowa; James Holmes, PhD, Principal Investigator — University of Iowa; Ruth L Chimenti, PT, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Health Care, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
All data that is necessary to validate primary outcomes and publications will be preserved and shared to allow other researchers the ability to reproduce the data and obtain additional findings that can advance the results. To ensure that other users can efficiently and accurately use the dataset, as well as to prevent misinterpretation or misuse, we will provide metadata and associated documentation. Information needed to understand the meaning of variable names and information about coding for missing data will be recorded in data dictionaries and readme files that will subsequently be shared alongside final datasets. Protocols, methods, statistical analyses, and any other relevant documentation derived from notes during data collection will be incorporated into readme files that will accompany the data when shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be available within 1 year of completing the study or upon publication, whichever occurs first. The data will remain available for at least 10 years. The primary outcome data and accompanying metadata will be deposited into an NIH Helping End Addiction Long-term (HEAL) compliant data repository.
Access Criteria: The primary outcome data and accompanying metadata will be deposited into an NIH Helping End Addiction Long-term (HEAL) compliant data repository. In accordance with International Committee of Medical Journal Editors (ICMJE), we will prepare the primary analysis datasets for review and reproducibility by peer-reviewed journals.
  Publications will be made available to the public using open access publishing, so that they become immediately available to the public. All publications will be accessible through PubMed, Google Scholar, and through open access.